CLINICAL TRIAL: NCT06869239
Title: Prediction of Response to PD-L1 Inhibitor After Chemoradiotherapy in Limited-Stage Small-Cell Lung Cancer Using Multi-omics-based Liquid Biopsy
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BRWEP2024W032150110
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Limited-stage Small Cell Lung Cancer (LS-SCLC)
Keywords: LS-SCLC; immunotherapy; liquid biopsy; high-dose radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Cisplatin; Carboplatin; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PD-L1 inhibitor after chemoradiotherapy: PD-L1 inhibitor maintenance following high-dose hyperfractionated simultaneous integrated boost radiotherapy concurrent chemotherapy in patients with limited-stage small cell lung cancer
  Interventions: Drug: Etoposide + cisplatin/carboplatin; Radiation: Thoracic radiotherapy; Radiation: Prophylactic cranial irradiation (PCI); Drug: PD-L1 inhibitor

INTERVENTIONS:
Drug: Etoposide + cisplatin/carboplatin — Four courses of intravenous cisplatin (75 mg/m² of body surface area on day 1 or divided into 3 days of each cycle) or carboplatin (area under the curve of 5 mg/mL per min on day 1 of each cycle) and intravenous etoposide (100 mg/m² of body surface area on days 1-3) every 3 weeks
Radiation: Thoracic radiotherapy — High-dose, accelerated, hyperfractionated, twice-daily thoracic radiotherapy (54 Gy in 30 fractions) concurrent with chemotherapy initiated at the beginning of cycles 1-3
Radiation: Prophylactic cranial irradiation (PCI) — PCI (25Gy in 10 fractions, once daily over two weeks) 3-4 weeks post-chemoradiotherapy for patients achieving PR or CR
Drug: PD-L1 inhibitor — Maintenance therapy with PD-L1 inhibitors (Durvalumab 1500 mg Q4W or Atezolizumab 1200 mg Q3W or Sugemalimab 1200 mg Q3W or Adebrelimab 1200 mg Q3W) post-PCI until disease progression, death, or intolerable toxicity, up to 2 years

SUMMARY:
This study aims to explore the efficacy and safety of immunotherapy (PD-L1 inhibitor) maintenance following high-dose hyperfractionated simultaneous integrated boost radiotherapy concurrent chemotherapy in patients with limited-stage small cell lung cancer (LS-SCLC). This study is a prospective observational study. Additionally, liquid biopsy technology will be employed to identify biomarkers that can predict the efficacy of PD-L1 inhibitor after chemoradiotherapy in LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years, male or female;
* 2. Histologically or cytologically confirmed limited-stage small cell lung cancer (LS-SCLC) (AJCC, 8th edition);
* 3. No more than 2 cycles of chemotherapy or no previous systemic therapy;
* 4. ECOG PS 0-1;
* 5. Measurable disease, as defined by RECIST v1.1 (tumor lesions long axis≥10mm, lymph nodes short axis ≥15mm);
* 6. Life expectancy ≥3 months;
* 7. Adequate pulmonary function;
* 8. Adequate hematologic and end-organ function, defined by the following criteria:

  1. Hematology

     * Hemoglobin (HGB) ≥90 g/L;
     * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L;
     * Platelet count (PLT) ≥ 100 x 10^9/L;
     * White blood cell count (WBC) ≥ 3.0 x 10^9/L;
  2. Serum chemistry

     * Serum albumin (ALB) ≥ 30 g/L;
     * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN;
     * Total bilirubin (TBIL) ≤1.5 ULN; Note: Patients diagnosed with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [mainly unconjugated bilirubin] without evidence of hemolysis or liver pathology) after consultation with their physician can be allowed;
     * Creatinine ≤ 1.5 ULN;
* 9. Women of childbearing age must have taken reliable contraceptive measures or undergone a negative pregnancy test (serum or urine) within 7 days prior to enrollment. Both men and women of childbearing age must agree to maintain adequate contraceptive measures throughout the study and for 6 months following the completion of treatment;
* 10. Patients must voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and actively cooperate with follow-up procedures.

Exclusion Criteria:

* 1. Histological mixture of SCLC and NSCLC components;
* 2. Extensive-stage SCLC;
* 3. Patients with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or those planned for transplantation;
* 4. Treatment with immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 14 days prior to the first dose of PD-L1 inhibitor, except for intranasal and inhaled corticosteroids or low-dose systemic steroids (i.e., ≤10 mg/day prednisolone or equivalent);
* 5. History of hypersensitivity to etoposide, cisplatin, PD-L1 antibody, or excipients in the formulation; or history of severe allergic reactions to other monoclonal antibodies;
* 6. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment;
* 7. Active or history of autoimmune disease or immune deficiency (including but not limited to autoimmune hepatitis, interstitial pneumonitis, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism);

Note:

* Patients with vitiligo or alopecia are eligible for this study;
* Patients with stable hypothyroidism undergoing hormone replacement therapy (e.g., Hashimoto's syndrome) are eligible for this study;

  * 8. Poorly controlled asthma despite systemic treatment, such as bronchodilators; Note: Patients with complete remission of asthma during childhood and no need for any intervention in adulthood can be allowed;
  * 9. Urinalysis shows proteinuria ≥ ++ or confirmed 24-hour urine protein ≥ 1.0g;
  * 10. Malignancies other than LS-SCLC, with the following exceptions:
* Adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix;
* Malignancy that has been treated with curative intent, with no known active disease for ≥5 years prior to the first dose of the study treatment, and with a low potential risk of recurrence;

  * 11. Human immunodeficiency virus (HIV) infection or known to have acquired immunodeficiency syndrome (AIDS);
  * 12. Significant cardiovascular disease within 6 months prior to enrollment, such as myocardial infarction, severe/unstable angina, New York Heart Association cardiac disease (class II or greater), poorly controlled arrhythmias (including QTcF interval >450 ms for males and >470 ms for females, with QTcF interval calculated using the Fridericia formula), and symptomatic congestive heart failure;
  * 13. Severe infections within 4 weeks prior to first dose of study treatment, including but not limited to infections requiring intravenous antibiotics, antifungal, or antiviral agents , or unexplained fever ≥38.5°C occurring during the screening period or before the first dose of the study treatment;
  * 14. Active tuberculosis, hepatitis B (HBV-DNA ≥ 500 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection of the assay), or co-infection with both hepatitis B and C;
  * 15. Treatment with any other investigational agent with therapeutic intent within 4 weeks prior to the first dose of the study treatment;
  * 16. History of abuse of psychotropic drugs or drug addiction;
  * 17. Patients with other severe physical or mental illnesses or abnormal laboratory test results that may increase the risk of participating in the study, or interfere with the study results, as well as those whom the investigator deems unsuitable for participation in the study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: LS-SCLC with PD-L1 inhibitor after Chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2028-01-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From enrollment to disease progression or death due to any cause, whichever occurs first, assessed up to 3 years.
  The time from enrollment to disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | The time from enrollment to death due to any cause, assessed up to 3 years.
  The time from enrollment to death due to any cause.
Objective response rate | Up to 3 years
  The percentage of participants who have a CR or a PR, as determined by investigators according to RECIST v1.1.
Disease control rate | Up to 3 years
  The percentage of participants who have a CR, a PR or a SD, as determined by investigators according to RECIST v1.1.
Incidence and severity of adverse events | From enrollment to 30 days after the end of study treatment.

OTHER OUTCOMES:
Blood biomarker analysis | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD related to article disclosure data
Supporting Information: Study Protocol
Time Frame: Available after publication
Access Criteria: Request by email to PI